CLINICAL TRIAL: NCT01038206
Title: Familias Unidas Stage III Study: Preventing Substance Abuse in Hispanic Youth
Brief Title: Familias Unidas: Preventing Substance Abuse in Hispanic Youth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DA025192-01A1
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Prevention; Family Function; Substance Use; Sexual Behavior
Keywords: prevention; HIV; drugs; smoking; Hispanic; Adolescent; Familias Unidas; Parent-Preadolescent Training; parent-centered; unsafe sexual behavior; efficacy; intervention
MeSH Terms: conditions — Substance-Related Disorders; Sexual Behavior; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Function Intervention (Experimental): Familias Unidas Intervention Program
  Interventions: Behavioral: Familias Unidas
- Treatment as Usual (No Intervention): The Public School system mandates that all high school students receive at least 5 lessons (55 minutes each) per year of HIV prevention.

INTERVENTIONS:
Behavioral: Familias Unidas — There will be 8 group sessions and 4 family visits. During the group sessions, the facilitator offers support for parents and gently corrects maladaptive interactions between parents and adolescents. During family visits, facilitators assist families in practicing skills and restructuring family interactions. The parent group sessions focus on parental investment in the adolescent's worlds (e.g., peer and school worlds), family communication, family support, behavior management/positive parenting, parental monitoring, adolescent substance use, and adolescent unsafe sex and HIV. Consistent with our prior Familias Unidas efficacy studies, all parent group sessions and all family visits will be conducted in Spanish and will take place in the evenings and on Saturdays at the school or at a community site that is preferred by the families.
  Arms: Family Function Intervention

SUMMARY:
The focus of this study will be to test the Familias Unidas Intervention program among Hispanic 8th graders in the Miami-Dade County Public School System. This study will contribute to the advancement of knowledge in both the scientific community and the Hispanic population in Miami-Dade County. It will shed light on whether and to what extent Familias Unidas is effective in preventing drug use and unsafe sexual behavior in Hispanic adolescents. To the scientific community, the investigators will disseminate our findings via peer-reviewed publications and presentations at scientific meetings.

The design for the proposed study is a randomized controlled trial. This design is considered the "gold standard" design when evaluating the efficacy of two (or more) treatment conditions. Participants for this study will be 744 Hispanic 8th grade adolescents and their parents recruited from 24 randomly selected middle schools in Miami Dade County that meet the school inclusion/exclusion criteria. A total of 12 schools (for a total of 372 Hispanic adolescents and their parents) will be randomized to Familias Unidas and a total of 12 schools (for a total of 372 Hispanic adolescents and their parents) will be randomized to the Community Practice.

DETAILED DESCRIPTION:
Substance use (including cigarette and illicit drug use) and HIV represent major public health problems facing America's youth (CDC, 2007; Johnston, O'Malley, Bachman, & Schulenberg, 2007). Hispanic adolescents report higher use across all drug categories (with the exception of amphetamines) and higher cigarette use than non-Hispanic White and African American adolescents (Johnston et al., 2007). Hispanic youth also engage in higher rates of unprotected sexual behavior at last sexual intercourse than non-Hispanic White and African American adolescents (CDC, 2007). Compared to non-Hispanic Whites, Hispanics are also disproportionately represented among HIV/AIDS cases, accounting for 18% if all such cases in the United States (CDC, 2006). These disparities are especially disconcerting because Hispanics are the largest and fastest growing minority group in the United States (Marotta & Garcia, 2003). Preventing substance use and HIV in Hispanic adolescents is therefore if vital importance.

Familias Unidas is delivered through family-centered, multi-parent groups that place parents in the change agent role and through family visits. Each parenting skill is discussed and role-played in parent-group sessions and is then enacted with the parent and the adolescent in a family visit. During the group sessions, the facilitator offers support for parents and gently corrects maladaptive interactions between parents and adolescents (during the group-session role plays, the role of adolescent is played by another parent). During family visits, facilitators assist families in practicing skills and restructuring family interactions. The parent group sessions focus on parental investment in the adolescent's worlds (e.g., peer and school worlds), family communication, family support, behavior management/positive parenting, parental monitoring, adolescent substance use, and adolescent unsafe sex and HIV. Consistent with our prior Familias Unidas efficacy studies, all parent group sessions and all family visits will be conducted in Spanish and will take place in the evenings and on Saturdays at the school or at a community site that is preferred by the families.

The proposed study will be guided by four aims. AIM 1 is to evaluate the effectiveness of Familias Unidas, relative to Community Practice (i.e., standard prevention services), in preventing illicit drug use in a community sample of Hispanic adolescents; AIM 2 is to evaluate the effectiveness of Familias Unidas, relative to Community Practice in preventing cigarette use in a community sample of Hispanic adolescents; AIM 3 is to evaluate the effectiveness of Familias Unidas, relative to Community Practice, in preventing unsafe sexual behavior in a community sample of Hispanic adolescents; and AIM 4 is to assess the extent to which family functioning mediates the effects of the intervention on illicit drug use, cigarette use, and unprotected sexual behavior.

Hypothesis 1. Familias Unidas will be more effective than Community Practice in reducing adolescent illicit drug use (defined as frequency of illicit drug use in the past 90 days) over time.

Hypothesis 1a. The effect of Familias Unidas on illicit drug use will be partially mediated by improvements in family functioning, defined as parental involvement, parental monitoring of peers, parent-adolescent communication, social support, and positive parenting.

Hypothesis 2. Familias Unidas will be more effective than Community Practice in reducing cigarette use (defined as frequency of cigarette use in the past 90 days) over time.

Hypothesis 2a. The effect of Familias Unidas on cigarette use will be partially mediated by improvements in family functioning, defined as parental involvement, parental monitoring of peers, parent-adolescent communication, family support, and positive parenting.

Hypothesis 3. Familias Unidas will be more effective than Community Practice in reducing unsafe sexual behavior (defined as unprotected sexual behavior at last sexual intercourse) over time.

Hypothesis 3a. The effect of Familias Unidas on unsafe sexual behavior will be partially mediated by improvement in family functioning, defined as parental involvement, parental monitoring of peers, parent-adolescent communication, family support, and positive parenting.

Inclusion/Exclusion criteria

a) Female and male adolescents of Hispanic origin, defined as self-identified Hispanic by the Primary caregiver.

(b) Adolescents attending 8th grade at baseline

(c) Adolescents living with an adult primary caregiver who is willing to participate

(d) At baseline, families must live within the catchment areas of the 24 participating middle schools

ELIGIBILITY:
Inclusion Criteria:

* Female and male adolescents of Hispanic immigrant origin, defined by the Primary caregiver as Self-identified Hispanic.
* Adolescents attending 8th grade at baseline
* Adolescents living with an adult primary caregiver who is willing to participate
* At baseline, families must live within the catchment areas of the 24 participating middle schools

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Substance use will be assessed using items extracted from the Monitoring the Future Study. | Three years
Adolescent unsafe sexual behavior will be measured using Jemmott, Jemmott, and Fong's (1998) 37-item Sexual Behavior instrument. | Three years

SECONDARY OUTCOMES:
Two subscales of the Parenting Practices: (a) extent of parental involvement (including involvement in school related activities) and (b) positive parenting will be used to assess parental investment. | Three years
The Family Relations Scale (6 items), completed by adolescent and parent, assess the amount of social support the adolescent receives from the parent | Three years
Parental investment in the adolescent will be assessed using (1) the Parenting Practices (2) the Family Relations scale | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, PhD, Principal Investigator — University of Miami
Locations (1):
- Center for Family Studies and Miami-Dade County Public Schools, Miami, Florida, United States

REFERENCES:
- [Derived] Lee TK, Estrada Y, Soares MH, Sanchez Ahumada M, Correa Molina M, Bahamon MM, Prado G. Efficacy of a Family-Based Intervention on Parent-Adolescent Discrepancies in Positive Parenting and Substance Use Among Hispanic Youth. J Adolesc Health. 2019 Apr;64(4):494-501. doi: 10.1016/j.jadohealth.2018.10.002. Epub 2018 Dec 1. PMID 30514652
- [Derived] Estrada Y, Lee TK, Huang S, Tapia MI, Velazquez MR, Martinez MJ, Pantin H, Ocasio MA, Vidot DC, Molleda L, Villamar J, Stepanenko BA, Brown CH, Prado G. Parent-Centered Prevention of Risky Behaviors Among Hispanic Youths in Florida. Am J Public Health. 2017 Apr;107(4):607-613. doi: 10.2105/AJPH.2017.303653. Epub 2017 Feb 16. PMID 28207330